CLINICAL TRIAL: NCT02791022
Title: A Multi-centre Population-based Study on the Incidence of Paroxysmal Atrial Fibrillation in Inpatient and Outpatient Cohorts in Singapore
Brief Title: Singapore Atrial Fibrillation Study
Acronym: SAFS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Changi General Hospital (Other); Singapore General Hospital (Other); National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/2309
Record Dates: First submitted 2016-05-30; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SPYDER ECG sensor

SUMMARY:
Atrial fibrillation is a common disease in the aging population that has severe implication if left untreated as it leads to embolic stroke and other embolic phenomenon. Embolic stroke in particular has severe implications to our community as the cost of care for such immobile patients can be extremely high. Atrial fibrillation typically begins as Paroxysmal atrial fibrillation (PAF), which makes early detection extremely difficult as the PAF may only occur transiently in the initial stages. Long term continuous ECG monitoring is currently required over weeks to detect early PAF. Current devices typically need to be implanted (loop recorders) to be sensitive enough to detect infrequent episodes of PAF. New generation ECG remote devices (non-invasive) are however now available that are wearable over long periods and can send data directly to a database for centralized collection and analysis of the data. The aim of this study will be to use such a device to evaluate the incidence of PAF in different population of patients, with each patient wearing and sending continuous ECG data for periods of a week or more to a central database, across several public hospitals in Singapore.

DETAILED DESCRIPTION:
The implications of PAF detection in an individual are huge to the individual and the community as it increases the risk of embolic stroke and other embolic phenomenon. Once detected, intervention can be taken to lower such an individual's clinical risk and decrease the clinical burden to the community. The lack of suitable tools and large population cohorts has led to a likely underestimation of PAF in various patient populations. This study will specifically address and characterize the different incidence on PAF in various patient populations and hence help to target at risk groups for earlier screening and intervention.

Patients with HF are more likely than the general population to develop AF. Conversely AF is also a strong independent risk factor for subsequent development of HF.

In Heart Failure (HF) patients, later development of AF was associated with increased mortality. Preexisting HF adversely affected survival in individuals with AF. Both HF with reduced ejection fraction (HFrEF) and Heart Failure with a Preserved Ejection Fraction (HFpEF) patients are at greater risk for AF. There is a direct relationship between functional state (as shown by the NYHA class) and prevalence of AF in patients with HF progressing from 4% in those who are NYHA class I to 40% in those who are NYHA class IV.

Acute HF decompensation in patients with prior HF is due to AF as a precipitant in 5.4% of cases in a single center study.

Knowing the true prevalence of AF in HF will allow us to plan for strategies to further reduce the clinical burden of HF.

ELIGIBILITY:
Inclusion Criteria:

1. Any male or female patient aged 21 years until 80 years old.
2. Not diagnosed to have atrial fibrillation
3. Patient must have sinus rhythm on 12 lead ECG prior to recruitment
4. Patient must be living in Singapore.
5. Ability to provide informed consent.
6. . Fulfill one or more of the risk factors stated below:

i) Hypertension

ii) Coronary arterial disease

iii) Ischemic heart disease

iv) Past history of congestive cardiac failure

v) Cerebrovascular accident

vi) Diabetes mellitus

Exclusion Criteria:

1. Known atrial fibrillation
2. Unable to use and manage a smartphone
3. Skin allergy to adhesive tape or plaster
4. Skin too hairy to apply device adhesive tape
5. Unable to comply with investigator's instructions and study protocols.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is 2500 inpatients and outpatients recruited from 4 medical institutions over a period of 3 years
  Power Calculation: This is a pilot study exploring the utility of employing a wearable device to detect the prevalence of PAF in the study populations.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Paroxysmal Atrial Fibrillation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chi Keong Ching, Principal Investigator — Singhealth Foundation
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No